CLINICAL TRIAL: NCT05486390
Title: EMPOWERing Patients With Chronic Diseases Through Smartphone App, Health Coaching and Shared Decision Making
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: SingHealth Polyclinics (Other); National University of Singapore (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202203-00046
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
Keywords: Nudge; Wearable; Behavioural change
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Nudge, health coaching and shared decision-making
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Nudge, health coaching and shared decision-making — The EMPOWER app aims to nudge the participant towards successful self-management of their diabetes condition by encouraging and reinforcing positive lifestyle behaviors in 3 main aspects - diet, physical activity, medication adherence. Notifications included content based on behavioural change technique including feedback on performance, positive reinforcement, and prompts to self-monitor. Each notification focused on a single behaviour (physical activity, medication adherence or diet).
  The participants in the intervention group will also interact with health coach throughout the study duration. In this study, the health coach will be responsible for the following roles :
  1. Goal setting and action plan
  2. After-visit summary
  A report card summarizing the lifestyle behaviour, goals will be made available to facilitate shared decision making.
  Arms: Intervention

SUMMARY:
Chronic diseases are the leading cause of deaths in Singapore. The rising prevalence in chronic diseases with age and Singapore's rapidly aging population calls for new models of care to effectively prevent the onset and delay the progression of these diseases. Advancement in medical technology has offered new innovations that aid healthcare systems in coping with the rapid rising in healthcare needs. These include mobile applications, wearable technologies and machine learning-derived personalized behaviorial interventions. The overall goal of the project is to improve health outcomes in chronic disease patients through delivering targeted nudges via mobile application and wearable to sustain behavioral change. Our overall objective is to design, develop, and evaluate an adaptive intervention platform on wearable devices and shared decision-making during consultations for patients with diabetes and hypertension. Our aim for this study is to assess the clinical effectiveness of real-time personalized educational and behavioural interventions delivered through wearable (Fitbit) and an integrative mobile application in improving patient glycaemic control measured using HbA1c over 9 months. Secondary outcomes will include change in systolic blood pressure, quality of life (QoL), patient activation, medication adherence, physical activity level, diet, direct healthcare cost and indirect healthcare cost over 9 months. We will conduct a randomized controlled trial among patients with comorbid diabetes and hypertension. This proposal aims to develop sustainable and cost-effective behavioural change among patients with comorbid diabetes and hypertension through patient empowerment and targeted chronic disease care.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21 years old and above
2. Have been diagnosed with diabetes at time of recruitment
3. Most recent glycated haemoglobin (HbA1c) ≥ 7.0%
4. Systolic blood pressure≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg on two or more prior visits, physician-diagnosed hypertension, or on antihypertensive medication
5. Physically able to exercise
6. Literate in English
7. Agreeable to be monitored by EMPOWER and/or Fitbit apps
8. Able to conform to monitoring schedule

Exclusion Criteria:

1. On bolus insulin treatment
2. Require assistance with basic activities of daily living (BADL)
3. Have planned major operation or surgical procedure within next 9 months
4. Cognitively impaired (scored ≥ 6 on the Abbreviated Mental Test)

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 9 months
  HbA1c over 9 months

SECONDARY OUTCOMES:
Systolic blood pressure | 9 months
  Systolic blood pressure over 9 months
Physical activity as measured by number of steps | 9 months
  Physical activity over 9 months
Physical activity as measured by moderate to vigorous active minutes | 9 months
  Physical activity over 9 months
Patient activation score as measured by patient activation measure | 9 months
  Difference in patient activation score between intervention and control over 9 months
Medication adherence as measured by Voils Scale | 9 months
  Difference in medication adherence between intervention and control over 9 months
Quality of life as measured by EQ-5D-5L | 9 months
  Difference in quality of life between intervention and control over 9 months
Healthcare cost | 9 months
  Healthcare cost over 9 months

CONTACTS AND LOCATIONS:
Locations (3):
- Singapore (3):
  - SingHealth Polyclinic (Bedok), Singapore
  - SingHealth Polyclinic (Punggol), Singapore
  - SingHealth Polyclinic (Tampines), Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwan YH, Yoon S, Tai BC, Tan CS, Phang JK, Tan WB, Tan NC, Tan CYL, Koot D, Quah YL, Teo HH, Low LL. Empowering patients with comorbid diabetes and hypertension through a multi-component intervention of mobile app, health coaching and shared decision-making: Protocol for an effectiveness-implementation of randomised controlled trial. PLoS One. 2024 Feb 26;19(2):e0296338. doi: 10.1371/journal.pone.0296338. eCollection 2024. PMID 38408067